CLINICAL TRIAL: NCT03841019
Title: Research on the Prediction of Clinical Response to Magnetic Seizure Therapy for Patients With Major Depression Episode
Brief Title: Predict MDE Outcomes After MST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201840269
Record Dates: First submitted 2019-01-17; First posted 2019-02-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Episode

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnetic seizure therapy (Experimental): 12 treatment sessions of MST, three times per week.
  Interventions: Device: Magpro X100 + Option
- electroconvulsive therapy (Active Comparator): 12 treatment sessions of ECT, three times per week.
  Interventions: Device: ThymatronSystem Ⅳ Electroconvulsive System

INTERVENTIONS:
Device: Magpro X100 + Option — In addition to treatment as usual (TAU), participants were supposed to receive twelve sessions of MST in four weeks (three sessions per week)
  Arms: magnetic seizure therapy
Device: ThymatronSystem Ⅳ Electroconvulsive System — In addition to treatment as usual (TAU), participants were supposed to receive twelve sessions of ECT in four weeks (three sessions per week)
  Arms: electroconvulsive therapy

SUMMARY:
This trial attempts to explore the treatment outcome of magnetic seizure therapy (MST) for major depressive episode. Half of the participants will receive MST, while the other half will receive electroconvulsive therapy (ECT).

DETAILED DESCRIPTION:
Magnetic seizure therapy (MST) is likely to be an alternative options to electroconvulsive therapy (ECT).

Widespread stimulation of cortical and subcortical regions is inevitable for ECT since the substantial impedance of the scalp and skull shuts most of the electrical stimulus away from the brain. Nevertheless, magnetic pulses are capable to focus the stimulus to a specific area of the brain because they can pass the scalp and skull without resistance. In Addition, electric current will penetrate into deeper structures, while magnetic stimulus are only capable to reach a depth of a few centimeters. As a consequence, MST are able to generate focus stimuli on superficial regions of the cortex while ECT can't, which may give MST the capability to produce comparable therapeutic benefits with the absence of apparent cognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of major depressive episode;
2. convulsive therapy clinically indicated, such as severe psychomotor excitement or retardation, attempts of suicide, being highly aggressive, pharmacotherapy intolerance, and ineffectiveness of antipsychotics;
3. the HAMD-17 ≥ 24;
4. informed consent in written form.

Exclusion Criteria:

1. primary diagnosis of other mental disorders;
2. severe physical diseases, such as stroke, heart failure, liver failure, neoplasm, and immune deficiency;
3. present with a laboratory abnormality that could impact on efficacy of treatments or safety of participants;
4. failure to respond to an adequate trial of ECT lifetime;
5. are pregnant or intend to get pregnant during the study;
6. Unremovable metal implants.
7. other conditions that investigators consider to be inappropriate to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
changes in the 17-item Hamilton Depression Rating Scale (HAMD-17) | At baseline and 4-week follow-up
  The HAMD-17 score ranges from 0 to 52. A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
changes in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | At baseline and 4-week follow-up
changes in the spectral power of the electroencephalogram (EEG) in square microvolt during resting state | At baseline and 4-week follow-up
changes in the spectral power of the electroencephalogram (EEG) in square microvolt during the auditory mismatch negativity task | At baseline and 4-week follow-up
changes in the spectral power of the electroencephalogram (EEG) in square microvolt during the facial recognition task. | At baseline and 4-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Sheng, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No